CLINICAL TRIAL: NCT04703556
Title: Recording and Modulation of Brain Activity Through Chronically Implanted Stimulation Electrodes in Patients With Parkinson's Disease
Brief Title: Recording and Modulation of Brain Activity Through Chronically Implanted Stimulation Electrodes
Acronym: PDNeuroGAIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol too complex for study population and difficulty to recruit participants with DBS and gait deficits
Sponsor: Jocelyne Bloch (Other)
Collaborators: Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Neurosurgeon, Professor in Neurosurgery, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBSgait2020
Record Dates: First submitted 2020-12-01; First posted 2021-01-11 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Gait and balance deficits; Deep brain stimulation; Neural sensing
MeSH Terms: conditions — Parkinson Disease | interventions — Equipment and Supplies; Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Single blinded study on patients with Parkinson's disease being treated with deep brain stimulation, who still experience severe therapy-resistant gait disorders.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Devices for deep brain stimulation — Effect of DBS parameters (amplitude, frequency) on gait and balance deficits, and their dynamical evolution over a pre-defined time

SUMMARY:
For decades, deep brain stimulation (DBS) therapies have been employed very successfully to alleviate segmental motor symptoms (tremor, brady-kinesia or rigidity) in patients with Parkinson's disease (PD). Unfortunately these therapies often fail to alleviate, or can even aggravate, axial deficits such gait and balance disorders. This is presumably due to the divergence in the dynamics of the circuits that control leg function, which are not well addressed with commonly employed stimulation protocols.

To date, patients still endure life-long debilitating gait difficulties that severely affect their everyday mobility, independence and quality of life.

In recent years, a handful of studies have proposed new paradigms, for instance using different stimulation parameters that are thought to be better suited for targeting the circuits that control lower limb function. Although promising, the resulting observations have been far from conclusive. As a result, the relevant approaches for therapeutic intervention remain unclear, and the underlying mechanisms largely unknown.

Advances on the use of implantable neuromodulation devices and of tech-nologies for monitoring whole-body movement currently allow to study locomotor deficits in ecological environments, enabling the recording and modulation of motor and neural signals while patients perform activities of daily living, chronically, wirelessly and in real time.

DETAILED DESCRIPTION:
This project seeks to leverage the latest technological innovations for monitoring and modulating motor and neural states chronically, in order to comprehensively characterize gait deficits in PD, and to clarify the improvements ushered in by varying DBS parameters.

The resulting observations will establish a rigorous understanding that will open new avenues for the design of evidence-based, clinically-relevant DBS strategies for locomotor deficits.

Advances on the use of neural implants for electrical neuromodulation of deep brain structures are opening the unique opportunity to probing the function of dysfunctional circuits in patients suffering from a variety of neurological disorders.

To date, acute experiments using deep brain stimulation (DBS) implants, either in intra-operative setups or shortly after surgery during so-called "externalization" phases, have widened our understan-ding of the neural signatures that underlie various motor and non-motor symptoms, and helped optimi-ze therapeutical parameters to better address such impairments.

For instance, DBS therapies in Parkinson's disease (PD) have been refined over the past decades based on experiments that synergistically (i) explored and uncovered readouts of movement perfor-mance in response to changing stimulation parameters, (ii) identified the underlying neural biomar-kers from recordings of local field potentials, and even (iii) tested closed-loop strategies able to adapt in real-time to ongoing patient-specific requirements.

These advances have mostly been applied to (and been successful for) improving motor signs of the upper-limb such as tremor, bradykinesia or rigidity, which exhibit fast dynamical responses to changes in neuromodulation (in the range of minutes), and which can be studied in the context of simple motor tasks using tethered technologies while patients are safely sitting or lying. These conditions have made it possible to tweak, tune and optimize parameters based on simple easily measurable readouts of motor dysfunction, and to record neural signals with minimal movement-related artefacts in the meantime.

Unfortunately, these straightforward experimental conditions do not apply to the study of axial motor signs, such as locomotion:

* First, gait deficits are multi-faceted and high dimensional: Impairments are not merely restricted to leg movements, but also critically affect lower- and upper-limb coordination, trunk and pelvis oscillations, posture and balance. Their characterization thus requires of multi-modal sensing technologies and analytical methods able to capture all these aspects concurrently.
* Second, the emergence of key deficits (e.g. freezing of gait) necessitates of behavioural tasks that are more physically demanding and potentially risky, often involving multiple repetitions of back-and-forth stepping over longer distances or in environments that resemble everyday life activities. Patients thus need to be in a stable medical condition, and technologies must allow recordings of motor and neural states to be performed wirelessly.
* Finally, the modulation of neural circuits controlling gait have considerably slower dynamics in response to changes in DBS (up to several hours10) than those controlling upper limb function, hence imposing that monitoring and tuning protocols are stretched in time to appropriately capture such changes.

These requirements critically put forward the need to study and devise novel therapies for gait deficits in the chronic state, using multi-modal technologies that can concurrently record neural and motor states remotely, in real-time and for long periods of time.

This project seeks to leverage the latest technological innovations for monitoring and modulating motor and neural states chronically, in order to comprehensively characterize gait deficits in PD while patients execute a range of activities of daily living, and to clarify the improvements brought in by varying DBS parameters.

In past years, a handful of studies have proposed new stimulation paradigms aimed to better target the neural circuits that control lower limb function during gait11. For instance strategies sought to combine varying DBS frequencies, or to target additional anatomical targets. They all highlighted promising, yet far-from-conclusive results. To date, the relevant approaches for therapeutic intervention remain unclear, and the underlying mechanisms largely unknown. Patients still endure life-long, debilitating gait difficulties that severely affect their everyday mobility and independence: they often feel insecure about leaving their homes due to the high risk of fall-related injuries, require personal assistance, and in general see their quality of life significantly diminished.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old or more
* Informed Consent as documented by signature
* Diagnosed with Parkinson's disease, and being treated with deep brain stimulation therapies.
* Exhibiting severe locomotor deficits
* Agree to comply in good faith with all conditions of the recordings.

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another investigational study in the preceding 30 days
* Previous enrolment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Changes in gait performance induced by DBS parameters | Measurement of performance is performed every 15 minutes up to 60 minutes for every condition.
  Improvements in performance will be evaluated using the results of the 10 meter test
Changes in gait performance induced by DBS parameters | Measurement of performance is performed every 15 minutes up to 60 minutes for every condition.
  Improvements in performance will be evaluated using the results of the stand-up and go test
Changes in gait performance induced by DBS parameters | Measurement of performance is performed every 15 minutes up to 60 minutes for every condition.
  Improvements in performance will be evaluated using the results of a test that measures the time to complete a path that includes straight walking and turning to induce (and measure the durations of) freezing of gait
Changes in gait quality induced by DBS parameters | Quality of gait patterns is performed during one walking recording, every 15 minutes up to 60 minutes for every condition.
  Quality in gait will compare the walking patterns of each patient with respect to healthy subjects : for that, multi-factorial analysis will be applied on recordings of kinematics (3D positions of body-joints recorded using a motion capture system). These multi-faceted signals are discretised per gait cycle, zscored, and their correlations extracted through Principal Component Analysis, which allows to identify key patterns being modulated with the therapy.
Changes in global motor scores induced by DBS parameters | UPDRS scores will be measured by an expert clinician every 15 minutes after each gait recording, up to 60 minutes per condition
  Unified Parkinson's Disease Rating Scores (UPDRS III)
Changes in brain dynamics induced by DBS parameters | Neural recordings will be performed prior to each UPDRS recording (every 15 minutes)
  Changes in neural signatures (STN LFP for patients implanted with an IPG that allows sensing, e.g. Percept PC) will be measured at rest, to extract their temporal evolution and their correlation with motor scores for each condition
Changes in brain dynamics induced by DBS parameters | Neural recordings will be performed prior to each UPDRS recording (2 minute recording every 15 minutes)
  Changes in neural signatures (EEG at rest) will be measured to extract temporal changes and their correlation with motor scores for each condition

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon completion of the study. The process is yet to be defined